CLINICAL TRIAL: NCT04972435
Title: Effect of Multifocal Intraocular Lens on Contrast Sensitivity in Primary Angle-Closure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Naris Kitnarong, Associate professor, Siriraj Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Naris001
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Primary Angle Closure Glaucoma; Primary Angle Glaucoma Closure Suspect; Senile Cataract
Keywords: primary angle closure; primary angle closure glaucoma; cataract surgery; contrast sensitivity; intraocular lens
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Contrast Sensitivity

STUDY DESIGN:
Intervention Model Description: Cataract patients with PAC or PACG who schedule for phacoemulsification with intraocular lens implantation. The patients must decide preoperatively to use multifocal IOL or monofocal IOL (patient preference) after receiving clear information about those 2 IOL models. Postoperatively, the contrast sensitivity (CS)will be measured with the same method. The postoperative CS were compared between groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifocal intraocular lens group (Experimental): Cataract patients with PAC or PACG who underwent phacoemulsification with multifocal intraocular lens implantation.
  Interventions: Diagnostic Test: Contrast sensitivity
- Monofocal intraocular lens group (Sham Comparator): Cataract patients with PAC or PACG who underwent phacoemulsification with monofocal intraocular lens implantation which are the standard IOL.
  Interventions: Diagnostic Test: Contrast sensitivity

INTERVENTIONS:
Diagnostic Test: Contrast sensitivity — All subjects performed the contrast sensitivity measurement preoperatively and one time at 2 months postoperatively.

SUMMARY:
This prospective study included patients with primary angle-closure (PAC or primary angle-closure glaucoma (PACG) and visually significant cataract. Phacoemulsification with multifocal intraocular lens (MIOL) or monofocal IOL (mIOL) (patient preference) was performed. Collected data included best-corrected distant visual acuity (BCVA), intraocular pressure (IOP), anterior chamber depth (ACD), and contrast sensitivity (CS) measured at spatial frequency 1.5, 3.0, 6.0, 12.0, and 18.0 cycles per degree (CPD) preoperatively, and at 2-6 months postoperatively. Preoperative and postoperative parameters were compared to evaluate the effect of MIOL on CS in eyes with PAC or PACG.

DETAILED DESCRIPTION:
This prospective non-randomized clinical study was conducted at the Department of Ophthalmology of the Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand during January 2014 to December 2015. The study protocol and informed consent procedures were both approved by our center's institutional review board (IRB) (approval number Si 384/2014). Each patient provided written informed consent prior to participation.

Primary angle closure was defined as an eye with invisible non-pigmented trabecular meshwork greater than 180 degrees and evidence of peripheral anterior synechiae on gonioscopy without glaucomatous optic disc appearance, glaucomatous pattern visual field damage, or history of increased IOP. Primary angle closure glaucoma was defined as an eye with invisible non-pigmented trabecular meshwork greater than 180 degrees on gonioscopy with glaucomatous optic damage (cup-to-disc ratio greater than 0.5 and/or localized neuro-retinal rim defect) and history of increased IOP raising. Patients with PACG must have been under good disease control, which was defined as IOP under 20 mmHg with 1 to 3 topical anti-glaucoma medications without deterioration of visual field, except generalized depression from cataract. Intra-ocular lens calculation was performed at the baseline visit using IOL Master. All patients received information about the advantages and disadvantages of MIOLs (Tecnis ZMB00 or Acrysof IQ Restore SN6AD1) and of mIOLs (Tecnis ZCB00 or Acrysof IQ SN60WF) before choosing the type of IOL that they individually preferred. Cataract surgery was performed by a single surgeon. Topical anesthesia was applied before standard phacoemulsification (2.2 mm temporal clear cornea incision and continuous curvilinear capsulorhexis) and IOL implantation into the capsular bag. Eyes with any intraoperative or postoperative complication were excluded.

Data specific to uncorrected and best-corrected distant visual acuities (UCVA and BCVA) in logMar, auto-refraction, slit-lamp ophthalmoscopic examination, intraocular pressure (IOP) measurement with Goldmann applanation tonometry, contrast sensitivity (CS), anterior chamber depth (ACD), central corneal thickness (CCT), and axial length (AL) were collected on the preoperative screening day, and at the 2 to 6-month postoperative follow-up. CS was measured under normal room light (photopic) conditions to evaluate patient quality of vision during the performance of their daily activities using a Functional Vision Analyzer. This test produces sine-wave gratings of different spatial frequencies. The absolute values of distance CS were obtained at five spatial frequencies (1.5, 3, 6, 12, and 18 cycles per degree; CPD). Visante® AS-OCT was used to determine CCT and ACD. ACD was defined as the distance between the corneal endothelium and the anterior surface of the crystalline lens (preoperative) or iris plane (postoperative). Axial length was obtained using IOL Master.

Comparisons of continuous data with normal distribution were made using Student's t-test for unpaired data, and using Mann-Whitney U test for non-normally distributed data. A p-value of less than 0.05 was defined as denoting statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Visually significant cataract patients aged >18 years with PAC or PACG who underwent prophylaxis peripheral iridotomy at least 2 months prior to participation.

Exclusion Criteria:

* Patients with preexisting glaucomatous visual field defect, except generalized depression
* Any other concurrent ocular diseases that could affect visual acuity, except cataract
* History of ocular inflammation or ocular surgery, except laser peripheral iridotomy, which is a routine procedure for treating PAC/PACG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Contrast sensitivity | Preoperative (on screening day)
  Contrast sensitivity at partial frequency 1.5, 3.0, 6.0, 12.0, and 18.0 cycles per degree (CPD)
Contrast sensitivity | At 2nd month postoperatively
  Contrast sensitivity at partial frequency 1.5, 3.0, 6.0, 12.0, and 18.0 cycles per degree (CPD)

SECONDARY OUTCOMES:
Visual acuity | Preoperative (on screening day)
  Visual acuity at distance in LogMar
Visual acuity | At 2nd month postoperatively
  Visual acuity at distance in LogMar
Anterior chamber depth | Preoperative (on screening day)
  Anterior chamber depth
Anterior chamber depth | At 2nd month postoperatively
  Anterior chamber depth

CONTACTS AND LOCATIONS:
Locations (1):
- Naris Kitnarong, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teichman JC, Ahmed II. Intraocular lens choices for patients with glaucoma. Curr Opin Ophthalmol. 2010 Mar;21(2):135-43. doi: 10.1097/ICU.0b013e3283365154. PMID 20040877
- [Result] Kim CY, Chung SH, Kim TI, Cho YJ, Yoon G, Seo KY. Comparison of higher-order aberration and contrast sensitivity in monofocal and multifocal intraocular lenses. Yonsei Med J. 2007 Aug 31;48(4):627-33. doi: 10.3349/ymj.2007.48.4.627. PMID 17722234
- [Result] Kumar BV, Phillips RP, Prasad S. Multifocal intraocular lenses in the setting of glaucoma. Curr Opin Ophthalmol. 2007 Feb;18(1):62-6. doi: 10.1097/ICU.0b013e328011d108. PMID 17159450
- [Result] Montes-Mico R, Alio JL. Distance and near contrast sensitivity function after multifocal intraocular lens implantation. J Cataract Refract Surg. 2003 Apr;29(4):703-11. doi: 10.1016/s0886-3350(02)01648-6. PMID 12686237